CLINICAL TRIAL: NCT01447056
Title: Most Closely HLA-Matched Allogeneic LMP1/2-Specific Cytotoxic T Lymphocytes for Treatment of Patients With Relapsed EBV-Associated Diseases
Brief Title: Most Closely HLA-Matched CTLs for Relapsed Epstein Barr Virus(EBV)-Associated Diseases
Acronym: MALTED
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Carlos Ramos, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-28361-MALTED; MALTED (Other: BCM)
Record Dates: First submitted 2011-08-12; First posted 2011-10-05 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Hodgkin Lymphoma; Non-Hodgkin Lymphoma; Lymphoproliferative Disorder; Nasopharyngeal Carcinoma; Leiomyosarcoma; Severe Chronic Active EBV (SCAEBV)
Keywords: Hodgkin lymphoma; Non-Hodgkin lymphoma; Lymphoproliferative disorder; Nasopharyngeal carcinoma; Leiomyosarcoma; EBV Cytotoxic T Lymphocytes
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoproliferative Disorders; Nasopharyngeal Carcinoma; Leiomyosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LMP Specific T cells (Experimental): LMP specific T cells will be given by intravenous injection over 1-10 minutes through either a peripheral or a central line and the IV flushed with saline. The volume of infusion will depend upon the concentration of the cells when frozen, the dose level, and the size of the patient.
  Interventions: Biological: LMP specific T cells

INTERVENTIONS:
Biological: LMP specific T cells — Three dose levels will be evaluated:
  Dose Level 1: 2×10^7 cells/m2; Dose Level 2: 1×10^8 cells/m2; Dose Level 3: 2×10^8 cells/m2
  If patients have a partial response or have stable disease they will be eligible to receive up to 5 further doses of CTLs, each of which will consist of the same number as their first injection.

SUMMARY:
Patients have a type of a lymph node cancer called lymphoma, a tumor of the nasal passages called nasopharyngeal carcinoma (NPC), a tumor of a particular type of muscle called leiomyosarcoma (LMS) or a condition called severe chronic active EBV (SCAEBV) syndrome. The disease has come back, may come back or has not gone away after treatment. This voluntary research study uses special immune system cells called LMP-specific cytotoxic T lymphocytes, a new experimental therapy.

Some patients with these diseases show evidence of infection with the virus that causes infectious mononucleosis (called Epstein-Barr virus, or EBV) before or at the time of their diagnosis. EBV is found in the cancer cells of up to half of the patients with lymphomas, and in some cases of NPC and LMS, suggesting that it may play a role in causing these diseases. Those cancer cells (as well as some B cells in SCAEBV) that are infected by EBV are able to hide from the body's immune system and escape destruction. We want to see if special white blood cells, called T cells, that have been trained to kill cells infected by EBV can survive in the blood and affect the tumor.

This treatment with specially trained T cells has had activity against these viruses when the cells are made from patients with those diseases (or, after bone marrow transplant, from the patient's transplant donor). However, sometimes it is not possible to grow these cells; other times, it may take 2 to 3 months to make the cells, which may be too long when one has an active tumor. We are therefore asking if subjects would like to participate in this study, which tests if blood cells from a donor that is a partial match with the subject (or the transplant donor) that have been grown in the way described above can survive in the blood and affect the disease.

These LMP-specific CTLs are an investigational product not approved by the Food and Drug Administration.

DETAILED DESCRIPTION:
First, we will search our cell bank to see if there is a CTL line that is a match with the subject and his/her donor. This matching is done using HLA type, which measures 6 proteins on the cell surface. If HLA type has not been previously checked, we will do a blood draw (half to one tablespoon) so that this can be done.

These CTL lines have been made at Baylor College of Medicine from donors for other transplant patients or other normal donors from the National Marrow Donor Program. All donors have been screened in the same way that we screen blood donors. When the CTL lines were made, blood was taken from the donors and used to grow T cells. To do this, we first grew a special type of cells called dendritic cells or monocytes and we put a specially produced human virus (adenovirus) that carries the LMP genes into the dendritic cells or monocytes. They were then used to stimulate T cells. This stimulation trained the T cells to kill cells with LMP on their surface.

We then grew these LMP specific CTLs by more stimulation with EBV infected cells (made from the same blood). We also put the adenovirus that carries the LMP genes into these EBV infected cells so that we increased the amount of LMP that these cells had. These EBV infected cells were treated with radiation so they could not grow. Once we made sufficient numbers of T cells, we tested them to make sure they kill cells with LMP on their surface and froze them.

To make sure that these cells won't attack the subject's tissues, we will also test the cells against his/her own cells, which we will grow in the laboratory.

If the level of circulating T-cells in the patient is relatively high, s/he will receive one treatment of cyclophosphamide. This drug will decrease the numbers of the patient's own T-cells before the investigators infuse the LMP-specific cytotoxic T-lymphocytes. If the patient is already receiving chemotherapy, this may not be needed.

The LMP specific CTLs will be thawed and injected IV over 1-10 minutes. Initially, one dose of T-cells will be given. If after the first dose, there is a reduction in the size of the patient's disease, they can receive up to five additional doses of the T-cells if they wish.

This is a dose escalation study, which means that the doses of cells will be increased as more patients are treated, as long as the lower doses are determined to be safe.

ELIGIBILITY:
INCLUSION CRITERIA:

SCREENING:

1. Any patient, regardless of age or sex, with one or more of the following EBV-positive or associated disorders, regardless of the histological subtype: - Hodgkin lymphoma - Non-Hodgkin lymphoma - Lymphoproliferative disorder - Nasopharyngeal carcinoma - Leiomyosarcoma - Severe chronic active EBV infection syndrome (SCAEBV), defined as high EBV viral load in plasma or PBMC (> 4000 genomes per ug PBMC DNA) and/or biopsy tissue positive for EBV
2. Karnofsky/Lansky score 50% or more.
3. Informed consent explained to and signed by patient or parent/guardian able to give informed consent and given a copy.

TREATMENT:

1. Any patient, regardless of age or sex, with one or more of the following EBV-positive or associated disorders, regardless of the histological subtype: - Hodgkin lymphoma - Non-Hodgkin lymphoma - Lymphoproliferative disorder - Nasopharyngeal carcinoma - Leiomyosarcoma - Severe chronic active EBV infection syndrome (SCAEBV), defined as high EBV viral load in plasma or PBMC (> 4000 genomes per ug PBMC DNA) and/or biopsy tissue positive for EBV
2. The disease needs to be in one of the following stages: - At diagnosis or in first relapse AND the patient is unable to receive conventional chemotherapy for his/her condition. - In second or subsequent relapse. - With residual disease after autologous, syngeneic or allogeneic HSCT.
3. Life expectancy 6 weeks or more.
4. Tumor tissue is positive for EBV.
5. Karnofsky/Lansky score 50% or more.
6. Bilirubin less than 3 times higher than the normal limits, AST less than 5 times higher than the normal limits, Hgb greater than 8.0 g/dL and serum creatinine less than 3 times higher than the normal limits.
7. Pulse oximetry of greater than 90% on room air.
8. If post allogeneic HSCT, patient must not have less than 50% donor chimerism in either peripheral blood or bone marrow.
9. Clinical status at enrollment to allow tapering of steroids to less than 0.5 mg/kg/day prednisone at time of treatment.
10. Informed consent explained to and signed by patient or parent/guardian able to give informed consent and given a copy.
11. Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 3 months after the study is concluded. The male partner should use a condom.

EXCLUSION CRITERIA:

SCREENING:

1. Known HIV positivity.

TREATMENT:

1. Currently receiving any investigational agents or have received any tumor vaccines within previous 4 weeks.
2. Active acute grade III-IV graft-versus-host disease.
3. Severe intercurrent infection.
4. Received alemtuzumab or other anti-T-cell antibody within 28 days.
5. HIV seropositivity.
6. Pregnancy (due to unknown effects of this therapy on a fetus) or lactation.
7. Tumor in a location where enlargement could cause airway obstruction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Patients with dose limiting toxicities after T-cell infusions | 6 weeks
  To determine the safety of intravenous injections of third-party, partially HLA- matched, allogeneic Epstein Barr Virus (EBV)-specific cytotoxic T-lymphocytes (CTL) in patients with severe chronic active EBV (SCAEBV) infection or EBV-associated Hodgkin or non-Hodgkin lymphomas (HL/NHL), other lymphoproliferative disorders (LPD) or other malignancies (leiomyosarcoma and nasopharyngeal carcinoma)

SECONDARY OUTCOMES:
Safety and response to a repeated dosage regimen | 5 years
  To obtain preliminary information on the safety and response to a repeated dosage regimen.
Analysis of immune function of CTLs | 5 years
  To determine the survival and the immune function of third-party allogeneic EBV-specific CTL lines
Number of patients with an EBV and/or disease response to the CTLs | 6 weeks
  To assess anti-EBV and anti-tumor effects of third-party partially HLA- matched allogeneic EBV-specific CTL lines.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Ramos, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas